CLINICAL TRIAL: NCT05414227
Title: Research on the Association of Gut Microbes and Their Metabolites With Post-stroke Depression
Brief Title: The Association of Gut Microbes and Their Metabolites With Post-stroke Depression
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The Affiliated Hospital of Xuzhou Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: XYFY2022-KL204
Record Dates: First submitted 2022-06-08; First posted 2022-06-10 (Actual); Last update posted 2022-06-10 (Actual); Status verified 2022-06

CONDITIONS: Acute Ischemic Stroke
Keywords: Gut flora; Acute Ischemic Stroke; Prognosis
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Faecal samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- PSD: Depressed as assessed by the Hamilton Depression Scale 3 months after stroke
- Non PSD: Nondepressed as assessed by the Hamilton Depression Scale 3 months after stroke

SUMMARY:
In this study, the clinical data of patients with AIS were collected, 16s RNA was used to detect the composition and diversity of intestinal flora, and flow cytometry and mass spectrometry were used to detect intestinal flora-related metabolites in plasma，to explore the influence of gut microbiota and its metabolites on stroke prognosis.

DETAILED DESCRIPTION:
In recent years, more and more studies have been conducted on the gut-brain axis, and gut microbes can affect the brain by regulating immune responses, metabolites, and neurotransmitters. The composition of gut microbiota may affect stroke prognosis, including focal neurological deficits, cognitive impairment, anxiety and depression, and fatigue. In this study, 16s RNA was used to detect the composition and diversity of intestinal flora, and flow cytometry and mass spectrometry were used to detect intestinal flora-related metabolites in plasma. The clinical data of patients were collected, including age, gender, and medical history, NIHSS, mRS, MMSE, Patient Health Questionnaire-9（PHQ9）, Social Support Rating Scale（SSRS）, laboratory and radiology results. The neurological recovery of the patients was assessed after 3 and 6 months, and the presence or absence of post-stroke depression（PSD） and post-stroke fatigue（PSF） was assessed by the Hamilton Depression Scale, the Fatigue Severity Scale（FSS） and the Multidimensional Fatigue Scale（MFS）. To evaluate the relationship between gut microbiota and its metabolites and stroke prognosis.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who suffered from acute ischemic stroke
2. Within 7 days of the onset
3. Signing the informed consent, willing and able to attend all study visits

Exclusion Criteria:

1. Severe aphasia，dysarthria, hearing loss，cognitive and consciousness impairment and unable to cooperate
2. Previous diagnosis of depression or other mental disorder or who had recently accepted antidepressants or antipsychotics
3. Gastrointestinal disease, and pregnant or lactating women
4. Serious systemic diseases including malignant tumors
5. Any antibiotics, probiotics or prebiotic treatment within 1 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with ischemic stroke within 7 days of onset
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-06-06 (Actual); Primary Completion 2023-02-28 (Estimated); Study Completion 2023-05-31 (Estimated)

PRIMARY OUTCOMES:
The PSD Assessed by Hamilton Rating Scale for Depression (HAMD-17) Score | 3 months
  Mild depression（HAMD-17 Score≥7，<17）, moderate depression（HAMD-17 Score≥17，<24）, major depression（HAMD-17 Score≥24）
The PSD Assessed by Hamilton Rating Scale for Depression (HAMD-17) Score | 6 months
  Mild depression（HAMD-17 Score≥7，<17）, moderate depression（HAMD-17 Score≥17，<24）, major depression（HAMD-17 Score≥24）
The PSF Assessed by Fatigue Severity Scale（FSS） | 3 months
  Fatigue（≥36）
The PSF Assessed by Fatigue Severity Scale（FSS） | 6 months
  Fatigue（FSS Score ≥36）
Functional Independence Assessed by Modified Rankin Scale (mRS）score | 3 months
  MRS score range from 0 to 6. Favourable outcome (mRS score≤2), worse outcome (mRS score>2), and death (mRS score = 6)
Functional Independence Assessed by Modified Rankin Scale (mRS）score | 6 months
  MRS score range from 0 to 6. Favourable outcome (mRS score≤2), worse outcome (mRS score>2), and death (mRS score = 6)

SECONDARY OUTCOMES:
Gut microbial composition and diversity | First stool after admission
  Results of fecal bacteria by 16s RNA sequencing
Serum metabolites of gut microbiota | 7 days within stroke onset
  Serum metabolites of gut microbiota from stool, detected by liquid chromatography-mass spectrometry (LC-MS) combined technique
Serum inflammatory cytokines | 7 days within stroke onset
  Inflammatory cytokines in blood，detected by flow cytometry

CONTACTS AND LOCATIONS:
Overall Officials: Chen Renguo, Master, Study Chair — The Affiliated Hospital of Xuzhou Medical University
Locations (1):
- The Affiliated Hospital of Xuzhou Medical University, Xuzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No